CLINICAL TRIAL: NCT01605929
Title: Clinical Evaluation of the Ultrasound-Guided Retroclavicular Brachial Plexus Block
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn before IRB approval
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kamen Vlassakov, Director of the Division of Regional and Orthopedic Anesthesia, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P000874
Record Dates: First submitted 2012-05-16; First posted 2012-05-25 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Anesthesia; Upper Extremity Injury
Keywords: Anesthetics, local/administration & dosage; Brachial Plexus/ultrasonography; Humans; Nerve Block/methods; Upper Extremity/surgery; Catheters, Indwelling; Anesthesia, Conduction/methods; Analgesia/methods; Nerve Block/adverse effects
MeSH Terms: conditions — Arm Injuries; Agnosia | interventions — Catheterization; Mepivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retroclavicular Brachial Plexus Block (Experimental)
  Interventions: Procedure: Retroclavicular Brachial Plexus Block and Catheter Insertion

INTERVENTIONS:
Procedure: Retroclavicular Brachial Plexus Block and Catheter Insertion — A Sonosite ultrasound machine will be used to visualize the nerve and needle simultaneously. A Braun 18 g 4 inch Touhy needle with markings will be inserted into the skin and advanced toward the nerve. Once the optimal location is determined under ultrasound visualization, the local anesthetic, mepivacaine, will be injected beside the nerves. The dose of drug will be mepivacaine 1.5%, 0.5 cc/kg (with a minimum 30 cc and maximum of 50 cc.) A Braun 20 g closed tip polyamide catheter will be inserted next to the nerve and left in place to allow for additional medication to be given postoperatively.
  Other Names: Carbocaine

SUMMARY:
The primary objective of this prospective, descriptive study is to evaluate the success rate of the retroclavicular brachial plexus block and catheter placement in 60 adult patients undergoing hand, wrist, or forearm surgery. The investigators will also evaluate any difficulties performing the procedure, the onset time and distribution of the block, incidence of adverse events, and patient's acceptance of the block.

DETAILED DESCRIPTION:
Nerve blocks are used by anesthesiologists as methods of pain control or to allow for painless surgery on a limb, rendering a general anesthetic for surgery unnecessary. Local anesthetic medication is injected through a needle next to a nerve, often using an ultrasound machine to visualize both the needle and nerve simultaneously. A catheter, a small plastic tube, can be inserted next to the nerve in order to provide pain relief for hours or days after surgery.

The nerves that provide sensation to the forearm, wrist and hand are the radial, median, ulnar, musculocutaneous and medial nerve of the forearm. These nerves originate from a network of nerve fibers that exit the spinal cord at the level of the neck. They are tightly bundled together, forming the brachial plexus, from the neck to just above the axilla, providing the anesthesiologist with many locations to perform a nerve block. One such block, known as the infraclavicular block, approaches the nerves just beneath the clavicle and has been performed for decades.

This study aims to examine a new technique to block the brachial plexus, performed at a similar level as the infraclavicular brachial plexus nerve block. The ultrasound-guided retroclavicular brachial plexus block has the potential advantages of being easier to perform, more successful, less painful for the patient, and a better pathway for catheter placement. It differs from the infraclavicular nerve block in that the needle is inserted above the clavicle rather than below it. In addition, it will allow the anesthesiologist to have another approach to the brachial plexus, which can be utilized if patients cannot have an infraclavicular block or any other brachial plexus block due to anatomical changes, or infection at the sight.

The retroclavicular brachial plexus block was first used in two patients at Brigham and Women's Hospital in whom the infraclavicular approach was contraindicated due to anatomical changes after surgery or trauma. This procedure has been found to be a reliable way to perform a brachial plexus nerve block and has become a routine procedure at Brigham and Women's Hospital for hand or forearm surgery over the past three years.

In reviewing the literature, a similar procedure was introduced by Hebbard and Royse in 2007, but no patient data was reported. By assessing the procedure in a prospective study, the investigators will be able to describe the technique, the success rate and any complications in the literature to allow other anesthesiologists to potentially incorporate this block into their repertoire.

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery of hand, wrist or forearm
* American Society of Anesthesiologists (ASA) physical status of I-II
* age greater than 18 years
* ability to provide written informed consent

Exclusion Criteria:

* clinically significant coagulopathy
* infection at the injection site
* abnormal anatomy at the block site
* allergy to amide anesthetics
* severe pulmonary pathology
* pre-existing motor or sensory deficits in the operative limb
* pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Success Rate | 20 minutes after nerve block completed
  Success rate will be defined as the number of patients with anesthesia or analgesia in all five nerves below the elbow (median, ulnar, radial, musculocutaneous, median nerve of the forearm).

SECONDARY OUTCOMES:
Motor Function | 20 minutes after nerve block completed
  Strength of muscles innervated by radial, median, ulnar, musculocutaneous, and axillary nerves
Complication of Procedure | From nerve block completion to patient's arrival in PACU, with an expected average duration of 3 hours
  Pneumothorax, Horner's syndrome, Symptomatic phrenic nerve palsy, Local anesthesia toxicity, block failure, catheter dislodgement.
Followup of Block Resolution | 48-96 hours post Retroclavicular Brachial Plexus Block
  Pain/Bruising/Infection at injection site, Unresolved paresthesias/weakness of operative arm, Preferences for Future Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kamen Vlassakov, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Vlassakov K, Janfaza D. Ultrasound-Guided Retroclavicular Approach to the Brachial Plexus Cords. Abstract, 33rd Annual Regional Anesthesia Meeting and Workshops, 2008.
- [Background] Vlassakov K, Brooks M, Islami-Manuchehry A, and Janfaza D. Our First Experience with the Novel Ultrasound-Guided Retroclavicular Block of the Brachial Plexus Cords in Patients with Normal Anatomy, Abstract, 34th Annual Regional Anesthesia Meeting and Workshops, 2009.
- [Background] Hebbard P, Royse C. Ultrasound guided posterior approach to the infraclavicular brachial plexus. Anaesthesia. 2007 May;62(5):539. doi: 10.1111/j.1365-2044.2007.05066.x. No abstract available. PMID 17448088